CLINICAL TRIAL: NCT04595045
Title: Effectiveness of Botulinum Toxin Type A Infiltrations in the Gait and Quality of Life in Adults With Spastic Lower Limb Paresis Secondary to Multiple Sclerosis
Brief Title: Botulinum Toxin in Patients With Spastic Lower Limb Paresis Associated With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aránzazu Vázquez Doce (Other)
Responsible Party: Sponsor-Investigator, Aránzazu Vázquez Doce, Principal Investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LINITOX
Record Dates: First submitted 2020-09-09; First posted 2020-10-20 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Botulinum toxin type A
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with spastic lower limb paresis (Experimental): patients with spastic lower limb paresis secondary to Multiple Sclerosis
  Interventions: Drug: Botulinum toxin type A infiltrations

INTERVENTIONS:
Drug: Botulinum toxin type A infiltrations — Echo-guided infiltration of botulinum toxin type A (Dysport®) in the lower limbs according to normal service practice

SUMMARY:
Spastic paraparesis is one of the most disabling functional deficits in the population with multiple sclerosis between 18 and 80 years of age and at any functional level. Infiltration with Botulinum Toxin is a clinical practice that has been carried out for years with clinical evidence of improvement in the patient's walking patterns and quality of life. We assume that the infiltration of this product can generate a direct benefit in the walking ability of these patients and secondarily improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance and signature of informed consent.
* Age between 18 and 80 years old, both included.
* Patients with relapsing remitting multiple sclerosis (RRMS), progressive secondary (SP) and primary progressive (PP), with spasticity resistant to usual treatment, either because of the severity of the spasticity or because of intolerance to side effects.
* Outpatients with spastic paraparesis that causes gait deficiency.
* Patients with an EDSS score between 2 and 6, both included.
* Patients with segmental involvement in MAS >1 in two or more muscle groups in the lower extremities.
* Absence of cognitive disability. Score less than 5 on the SPMSQ scale of Pfeiffer.
* Possibility of carrying out the treatment (method of administration, scheduled visits) and scales correctly.
* Women of childbearing potential should use an effective contraceptive method (hormonal contraceptives, intrauterine device, condom) or refrain from having sex in order not to get pregnant. A woman is considered to be fertile after menarche and to become postmenopausal, unless she has undergone a permanent sterilization procedure (hysterectomy, salpingectomy, bilateral oophorectomy). A postmenopausal state is defined as absence of menstruation for 12 months without an alternative medical cause.

Exclusion Criteria:

* Psychiatric illness that hinders participation in the trial.
* Comorbidity that threatens the patient's life in the short term (severe liver disease, cardiovascular disease, etc.).
* Osteoarticular disorder that prevents physical activity.
* Pregnancy or lactation.
* Lack of primary or secondary response to any type of Botulinum Toxin for the treatment of MS previously detected.
* Sensitivity to Botulinum Toxin or to any excipient.
* Any medical condition that, in the opinion of the investigator, may compromise compliance with the objectives and / or procedures of this protocol or preclude the administration of Botulinum Toxin.
* Changes in the treatment regimen of any drug that directly or indirectly interferes with neuromuscular function within 4 weeks before the start of the study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Effectiveness of repeated Botulinum Toxin infiltrations using objective results obtained by the clinician (Six Minutes Walking Test - 6MWT). | 12 months
  To assess the effectiveness of repeated Botulinum Toxin infiltrations on gait in patients with Multiple Sclerosis who presented limb spasticity less than 4 weeks after infiltration and its maintenance over time at 12 months, using objective results obtained by the clinician (Six Minutes Walking Test - 6MWT). Higher scores mean a better outcome.
Effectiveness of repeated Botulinum Toxin infiltrations using results reported by the patient (Twelve item Multiple Sclerosis Walking Scale - MSWS-12). | 12 months
  To assess the effectiveness of repeated Botulinum Toxin infiltrations on gait in patients with Multiple Sclerosis who presented limb spasticity less than 4 weeks after infiltration and its maintenance over time at 12 months, using results reported by the patient (Twelve item Multiple Sclerosis Walking Scale - MSWS-12). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Evaluation of spasticity using Modified Ashworth Spasticity scale (MAS scale). | 12 months
  Evaluation of spasticity using Modified Ashworth Spasticity scale (MAS scale). Higher scores mean a worse outcome.
Evaluation of disability using Expanded Disability Status Scale de Kurtzke (EDSS scale). | 12 months
  Evaluation of disability using Expanded Disability Status Scale de Kurtzke (EDSS scale). Higher scores mean a worse outcome.
Evaluation of the quality of life after the use of botulinum toxin type A using Multiple Sclerosis Quality of Life 54 (MSQoL-54). | 12 months
  Evaluation of the quality of life after the use of botulinum toxin type A using Multiple Sclerosis Quality of Life 54 (MSQoL-54). Higher scores mean a better outcome.
Assessment of medium and long-term objectives using Goal Attainment Scaling (GAS scale). | 12 months
  Assessment of medium and long-term objectives using Goal Attainment Scaling (GAS scale). Higher scores mean a better outcome.
Number of adverse events. | 12 months
  Number of adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de la Princesa, Madrid